CLINICAL TRIAL: NCT00529620
Title: Randomized Trial of Effectiveness and Acceptability of Three Alternative Regimens for Malaria Seasonal Intermittent Preventive Treatment in Senegal
Brief Title: Three Alternative Drug Regimens for Malaria Seasonal Preventive Treatment in Senegal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Cheikh Anta Diop University, Senegal (Other)
Responsible Party: Dr Badara Cisse, University of Dakar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5184
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Malaria
Keywords: Malaria; IPT; preventive treatment
MeSH Terms: conditions — Malaria | interventions — Amodiaquine; artenimol; piperaquine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): sulfalene pyrimethamine plus amodiaquine
  Interventions: Drug: sulfalene-pyrimethamine plus amodiaquine
- 2 (Active Comparator): dihydroartemisinin piperaquine
  Interventions: Drug: dihydroartemisinin plus piperaquine
- 3 (Active Comparator): sulfadoxine-pyrimethamine plus piperaquine
  Interventions: Drug: sulfadoxine pyrimethamine plus piperaquine

INTERVENTIONS:
Drug: sulfalene-pyrimethamine plus amodiaquine — Monthly treatments during the malaria transmission season
  Other Names: Dualkin
  Arms: 1
Drug: dihydroartemisinin plus piperaquine — Monthly treatments during the transmission season
  Other Names: Duo cotexcin
  Arms: 2
Drug: sulfadoxine pyrimethamine plus piperaquine — Monthly treatments during the malaria transmission season
  Other Names: sulfadoxine pyrimethamine; piperaquine phosphate
  Arms: 3

SUMMARY:
The purpose of this trial is to compare the acceptability, efficacy and safety of three alternative drug regimens for use for seasonal Intermittent Preventive Treatment to prevent malaria in children. Children aged 2 months to 5 years will be randomized to receive IPT with one of three regimens during the transmission season: sulfadoxine-pyrimethamine (SP) plus amodiaquine, show to be highly effective for IPT in a recent trial; SP plus piperaquine, used for malaria prophylaxis in China for many years; or Duocotexcin (a combination of piperaquine with an artemisinin).

DETAILED DESCRIPTION:
In areas of seasonal malaria transmission the burden of severe disease and mortality due to malaria is mainly among children under 5 years of age. Intermittent preventive treatment (IPT) with antimalarial drugs given to all children once a month during the transmission season is a promising new strategy for malaria prevention. Seasonal IPT with sulfadoxine-pyrimethamine (SP) and one dose of artesunate resulted in a 90% reduction in incidence of clinical malaria in a recent trial in Senegal (Cisse et al., Lancet 2006). An important consideration is the possible impact of seasonal IPT on the emergence and spread of drug resistant parasite genotypes, the choice of drug regimen is therefore critical. A second trial in Senegal showed that a combination of two non-artemisinin drugs with relatively long half lives (SP and amodiaquine (AQ) over three days) was more effective than SP with artesunate and more effective than AQ with artesunate, in preventing malaria; and very few children developed parasitaemia, so that the potential for drug resistant genotypes to emerge and spread was low. Although SP+AQ was more efficacious than the artemisinin-containing regimens tested, it was associated with a higher frequency of adverse events, especially vomiting, and AQ has a bitter unpleasant taste, and therefore we have concerns about the acceptability of AQ for widespread use for IPT. It is important to select a drug regimen that is not only effective but safe and acceptable to the community. Each treatment is a 3-dose regimen over 3 days, the first dose will be supervised and the other 2 doses given by the mother or carer. One month after each treatment round, children will be visited at home to check for malaria symptoms, children with fever or a history of fever in the last 48 hours will be asked to give a finger prick blood sample for malaria diagnosis. One month after the last treatment all children will be asked to give a finger prick blood sample for parasitology and haemoglobin, axillary temperature will be measured. The child's carer will be interviewed about compliance and adverse events. The endpoints will be the cumulative incidence of malaria, the proportion of children experiencing moderate and severe adverse events, compliance with and acceptability of the regimen, the prevalence of parasitaemia, and the proportion of children carrying parasite genotypes associated with resistance to sulfadoxine or pyrimethamine at the end of the transmission season. Since acceptability is difficult to assess in the formal setting of a trial, and because the method of delivery may affect compliance and acceptability, drug treatments will be delivered by community workers replicating the conditions under IPT would be delivered routinely in Senegal. Treatments will be administered at home by local community workers, each worker covering a circuit of approximately 60-80 children. The community worker circuit will be the unit of randomization, for simplicity in the field to minimise allocation errors, and to avoid contamination due to sharing of tablets within a household.

ELIGIBILITY:
Inclusion Criteria:

* age 2 to 59 months in September 2007

Exclusion Criteria:

* history of allergy to study drugs

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1833 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Incidence of malaria | Four months

SECONDARY OUTCOMES:
Adverse events reported by the mother: vomiting, headache, fever, nausea, diarrhea | within 4 days of the start treatment
Prevalence of P.falciparum parasitaemia | Measured by microscopy 1 month after the last treatment, in December
Haemoglobin concentration | Measured 1 month after the last treatment, in December
The proportion of children carrying P.falciparum genotypes associated with resistance to sulfadoxine and pyrimethamine | Measured in December
Compliance with the treatment regimen | Recorded 4 days after the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Badara Cisse, PhD, Principal Investigator — Universite Cheikh Anta Diop; Paul J Milligan, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Departement de Parasitologie et Mycologie, Universite Cheikh Anta Diop, Dakar, Senegal

REFERENCES:
- [Derived] Cisse B, Cairns M, Faye E, NDiaye O, Faye B, Cames C, Cheng Y, NDiaye M, Lo AC, Simondon K, Trape JF, Faye O, NDiaye JL, Gaye O, Greenwood B, Milligan P. Randomized trial of piperaquine with sulfadoxine-pyrimethamine or dihydroartemisinin for malaria intermittent preventive treatment in children. PLoS One. 2009 Sep 28;4(9):e7164. doi: 10.1371/journal.pone.0007164. PMID 19784374